CLINICAL TRIAL: NCT03288610
Title: Prognostic Value of Copeptin Level Before Cardiac Surgery and Involvement in Systemic Inflammatory Response Syndrome After Cardiopulmonary Bypass
Brief Title: Prediction of Inflammatory Response and Hypotensive Syndrome After Cardiac Surgery by Preoperative Copeptin Level
Acronym: MicorSIRS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 9754
Record Dates: First submitted 2017-05-09; First posted 2017-09-20 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-05

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS); Postoperative Vasodilation Syndrome; Stress Response; Cardiac Surgery Prognosis; Tissue Oxygenation and Post-ischemic Response
Keywords: Copeptin; Vasopressin; Microcirculation; Inflammation; Vasodilation; Cardiopulmonary bypass
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Fractures, Stress; Diabetes Insipidus; Inflammation; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma: preoperative, ICU admission at POD0 and POD1 samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- With inflammatory response: Patients with postoperative inflammatory response as defined by the occurrence of severe SIRS and/or postoperative vasodilation syndrome.
  Severe SIRS is defined by meeting at least 2 SIRS criteria during 6 consecutive hours or at least 3 SIRS criterias. Classical SIRS criteria include: temperature >38,3 or <36°C, heart rate >90/min, respiratory rate >20/min or PaCO2 <32mmHg, GB>12000 ou <4000 c/mm3.
  Postoperative vasodilation syndrome is defined by the need of continuous infusion of norepinephrine (whatever the dose) to maintain the mean arterial pressure above 60 mmHg associated to a cardiac index above or egal to 2.2 L/min/m2.
  Patients without postoperative severe SIRS and without postoperative vasodilation syndrome
  Interventions: Diagnostic Test: Preoperative copeptin level

INTERVENTIONS:
Diagnostic Test: Preoperative copeptin level — Measure of plasmatic copeptin from preoperative samples retained in a biorepository. Physicians are blinded to the result.
  Other Names: Biomarker of vasopressin secretion; Systemic Inflammatory Response Syndrome (SIRS); Postoperative vasodilation syndrome; Stress response

SUMMARY:
The purpose of this study is to find a preoperative biomarker before cardiac surgery with cardiopulmonary bypass related to severe postoperative inflammatory response and circulatory complications. The investigators hypothesize that an increase of the preoperative stimulation of vasopressinergic system (in response to acute or chronic conditions) could lead to a microcirculatory dysfunction and favor the occurrence of vasodilatation during and after CPB and increase the symptoms of an inflammatory response after CPB. By defining a high risk population, a targeted strategy of monitoring and early or preventive treatment could improve postoperative prognosis.

DETAILED DESCRIPTION:
The occurrence of a severe systemic inflammatory response syndrome (SIRS) after elective cardiac surgery with cardiopulmonary bypass (CPB) is estimated at about 20% of cases and is characterized by hemodynamic changes (tachycardia, hypotension, hypovolemia). It is also responsible for vasodilation with impaired microcirculation involving increased morbidity and mortality associated with organ dysfunction and the risk of bacterial translocation. However, the participation of vasopressinergic system in the functional impairment of microcirculation is unclear.

Copeptin is considered a marker of vasopressin secretion, deriving from the same precursor, being more stable and easy to dose. In a previous study of 64 patients with CPB, the investigators have shown that high copeptin preoperative levels are associated with the occurrence of vasodilatation syndrome after cardiac surgery (incidence 15%) with a relative deficiency of postoperative vasopressin.

Microcirculatory alterations can be explored through the study of tissue oxygenation by NIRS (StO2) at rest and in response to a hypoxic challenge (provided by brief vascular occlusion). In septic shock, altered recovery slopes of tissue oxygenation are associated with poor prognosis. The investigators could find similar impact on prognosis in cardiogenic shock if first hours of care did not improve this recovery slope.

The investigators hypothesize that an increase of the preoperative stimulation of vasopressinergic system (in response to acute or chronic conditions) could favor the occurrence of vasodilatation during and after CPB and increase the symptoms of an inflammatory response after CPB. The involvement of vasopressin in microcirculatory dysfunction is unknown.

This is a validation study of a predictive test for pathophysiology and prognosis. This study will be monocentric, prospective and observational in routine care.

The main end point of the study is to predict the onset of severe SIRS or postoperative vasodilation syndrome after CPB by the preoperative plasma copeptin level in a cardiac surgery population.

The secondary objectives are to assess the incidences of microcirculatory dysfunction, shock and organs failure after CPB, to determine the postoperative copeptin kinetics for patients with severe SIRS, to evaluate the prognosis with the ICU length of stay and D28 mortality.

Data are recorded prospectively on a paper case report form by ICU physicians in charge of the patients on the basis of clinical observation and electronic medical records. Quality assurance, monitoring and auditing are provided by the study promotor. Data will be checked by the main investigator to assess the accuracy and completeness of entered data into the CRF.

Patients are recruited during the preoperative period after screening of inclusion and exclusion criteria, delivering information and obtaining written consent.

Considering an expected sensitivity for predicting SIRS by preoperative copeptin on the order of 80%, the number of cases (subjects with severe SIRS) to be included for obtaining an estimate of the sensitivity with a lower limit of 95% to 55% is placed in 42 cases. Considering an incidence of severe SIRS at 20%, the total number of patients to be included in the study is 200. In our center the investigators perform 700 CPB / year, 70% met the criteria for inclusion.

For the primary objective, the predictive performance of preoperative copeptin for the occurrence of post-CPB severe SIRS will be evaluated by the construction of a ROC curve with finding an optimal threshold maximizing sensitivity and specificity (calculation of the Youden index) to be then estimated with their 95% confidence interval.

Regarding the secondary objectives, copeptin levels will be compared according to the presence of postoperative microcirculatory dysfunction, hemodynamic failure, organ dysfunction and preoperative factors using a reduced gap test. Univariate and multivariate analysis using linear regressions will be carried out to find the preoperative factors associated significantly and independently to high copeptin level. The postoperative kinetics of copeptin will be modeled using mixed linear regressions with an intercept +/- a random slope and taking into account the intra-individual correlation of the assays. The prognostic value of preoperative copeptin and postoperative StO2 recovery slope on D28 mortality will be analyzed using the ROC curve, determination of an optimal threshold using the Youden index and then calculating Sensitivity and specificity with their 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Scheduled time of at least 24 hours
* Cardiopulmonary bypass

Exclusion Criteria:

* Urgent surgery within 24 hours of hospital admission
* Chronic renal failure with preoperative glomerular filtration rate below 45 ml/min
* Ongoing sepsis (ie uncontrolled endocarditis)
* Immunosuppressive therapy (solid organ transplant recipient)
* Previously included in this study

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized and scheduled for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Preoperative copeptin level | Preoperative 24 hours
  Plasmatic copeptine will be measured from routine blood sample on heparinazed tubes. The biological assay will be performed by Time-Resolved Amplified Cryptate Emission on automate Kryptor Compact plus (ThermoFisher, Clichy, France). A level above the 97° percentile of referent population will be considered pathological.

SECONDARY OUTCOMES:
Postoperative microcirculatory impairment | Within 2h of admission in intensive care unit, before weaning of sedation and mechanical ventilation
  Tissue oxygen saturation (STO2) measured at the thenar eminence by NIRS (Inspectra 650, Hutchinson Technologies) with application of a 3 min vascular occlusion test to measure the occlusion slope, the recovery slope and the hyperemic rebound. Microcirculatory dysfunction is defined by a recovery slope below 3%/s.
Occurrence of SIRS using classical definition | First postoperative 24 hours
  SIRS is classically defined when 2 of the following criteria are met together: temperature >38,3 or <36°C, heart rate >90/min, respiratory rate >20/min or PaCO2 <32mmHg, GB>12000 ou <4000 c/mm3.
Postoperative hemodynamical impairment | First postoperative 24 hours
  Occurrence of
  * A postoperative vasodilation syndrome defined by the need of continuous infusion of norepinephrine (whatever the dose) to maintain the mean arterial pressure above 60 mmHg associated to a cardiac index above or egal to 2.2 L/min/m2
  * a postoperative low cardiac output syndrome defined by cardiac index below 2.2 L/min/m2 without hypovolemia,
  * a tissue hypoxia assessed by 2 consecutive lactate level above 2.2 mmol/l,
  * an hemorrhagic shock or
  * a septic shock.
Perioperative copeptin kinetics | 24 hours before the operation until admission intensive care unit
  Plasmatic copeptin will be measured from routine blood sample on heparinized tubes. The biological assay will be performed by Time-Resolved Amplified Cryptate Emission on automate Kryptor Compact plus (ThermoFisher, Clichy, France). A level above the 97° percentile of referent population will be considered pathological.
Perioperative copeptin kinetics | postoperative day
  Plasmatic copeptin will be measured from routine blood sample on heparinized tubes. The biological assay will be performed by Time-Resolved Amplified Cryptate Emission on automate Kryptor Compact plus (ThermoFisher, Clichy, France). A level above the 97° percentile of referent population will be considered pathological.
Global organs dysfunction | First postoperative 24 hours
  Assessed by the Sequencial Organ Failure Assessment (SOFA) score calculated at the postoperative day
Lengh of mechanical ventilation | Up to 28 days
  Length (hours) of postoperative invasive mechanical ventilation
Acute kidney injury | Up to 28 days
  Defined and classified according to KDIGO criteria
Renal replacement therapy | Up to 28 days
  Incidence of patients requiring renal replacement therapy in ICU due to postoperative acute kidney injury
Intensive Care Unit stay | through study completion, an average of 3 month
  Length (days) of postoperative intensive care unit stay
Hospital stay | through study completion, an average of 3 month
  Length (days) of postoperative hospital stay before current care ward discharge (excluding rehabilitation time)
Intensive Care Unit mortality rate | Up to 28 days
  Intensive care unit mortality rate : death before ICU discharge
Day 28 mortality rate | Up to 28 days
  Overall mortality rate at 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gaudard, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Department of critical care, Arnaud de Villeneuve Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacCallum NS, Finney SJ, Gordon SE, Quinlan GJ, Evans TW. Modified criteria for the systemic inflammatory response syndrome improves their utility following cardiac surgery. Chest. 2014 Jun;145(6):1197-1203. doi: 10.1378/chest.13-1023. PMID 24576975
- [Result] Colson PH, Bernard C, Struck J, Morgenthaler NG, Albat B, Guillon G. Post cardiac surgery vasoplegia is associated with high preoperative copeptin plasma concentration. Crit Care. 2011;15(5):R255. doi: 10.1186/cc10516. Epub 2011 Oct 25. PMID 22026977